CLINICAL TRIAL: NCT05335109
Title: Neuroprotective Effects of Xenon Treatment in Patients with Cerebral Infarction: Randomized Single-blinded Placebo-controlled Trial
Brief Title: Neuroprotective Effects of Xenon Treatment in Patients with Cerebral Infarction
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Negovsky Reanimatology Research Institute (Other Government)
Responsible Party: Principal Investigator, Oleg A. Grebenchikov, The head of the laboratory in the Negovsky Reanimatology Research Institute, Negovsky Reanimatology Research Institute
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: NEXT
Record Dates: First submitted 2022-04-12; First posted 2022-04-19 (Actual); Last update posted 2024-10-03 (Actual); Status verified 2024-10

CONDITIONS: Ischemic Stroke
Keywords: Ischemic stroke; Xenon; Organ protection; Critical care
MeSH Terms: conditions — Ischemic Stroke | interventions — Xenon

STUDY DESIGN:
Who Masked: Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Xenon (Experimental)
  Interventions: Drug: Xenon
- Oxygen (Placebo Comparator)
  Interventions: Drug: Oxygen 30 %

INTERVENTIONS:
Drug: Xenon — Xenon is injected into the body by inhalation in the form of xenon-oxygen mixtures, in which the concentration of xenon is 30%, and oxygen is 30%.
  Xenon inhalation is carried out for 30 min daily for 3 days.
  Arms: Xenon
Drug: Oxygen 30 % — Oxygen-air mixture is injected into the body by inhalation. The oxygen concentration is 30%.
  Inhalation of oxygen-air mixture is carried out for 30 min daily for 3 days
  Arms: Oxygen

SUMMARY:
In the Russian Federation, ischemic cerebral infarction is recorded annually in more than 450,000 people. It is the second most common cause of death after coronary heart disease.

The 30-day mortality rate after an ischemic cerebral infarction is more than 25%, and during the following year about half of the patients die. To date, all candidate neuroprotective drugs tested in various clinical trials have demonstrated insufficient efficacy . Therefore, the development of new approaches to the treatment of severe brain injuries of various etiologies is one of the most important tasks of critical condition medicine.

Brain damage due to stroke triggers a number of pathophysiological reactions, which are based on the accumulation of glutamate with the development of excitotoxicity. The effect of glutamate on NMDA receptors is one of the main factors of neurodegenerative disorders.

Xenon is an anesthetic whose neuroprotective properties have been shown in many experimental studies. Хenon inhalation after ischemia and reperfusion suppresses ischemic brain damage and tPA-induced cerebral hemorrhages, and damage to the blood-brain barrier.

The most interesting is a randomized controlled trial performed by R. Laitio et al. (2016), in which the use of xenon in combination with hypothermia in clinical practice was studied for the first time. In patients who have undergone community-acquired cardiac arrest, xenon inhalation at a concentration of 40 vol.% within 24 hours in combination with hypothermia, led to less damage to the white matter of the brain than with patients using hypothermia alone. The 6-month mortality rate was 27% in the xenon and hypothermia group and 35% in the hypothermia group.

It is important to note that today, despite a large pool of convincing preclinical studies proving the neuroprotective properties of xenon, there is not a single clinical study of its use in ischemic stroke.

Therefore, the research objectives is to determine whether the strategy of using xenon-oxygen mixture inhalation is better than oxygen-air mixture inhalation with respect to the change in scores on the NIHSS, Rankin and Glasgow coma scales on day 7, the duration of stay in the ICU and the frequency of nosocomial pneumonia.

DETAILED DESCRIPTION:
In the Russian Federation, ischemic cerebral infarction is recorded annually in more than 450,000 people. It is the second most common cause of death after coronary heart disease.

The 30-day mortality rate after an ischemic cerebral infarction is more than 25%, and during the following year about half of the patients die, which is more than 200,000 people. The consequences of stroke belong to the first place among the causes of primary disability. No more than 15% of those who have suffered a stroke return to work or fully perform their previous household duties, and the rest, due to disability, need lifelong medical and social rehabilitation. To date, all candidate neuroprotective drugs tested in various clinical trials have demonstrated insufficient efficacy . Therefore, the development of new approaches to the treatment of severe brain injuries of various etiologies is one of the most important tasks of critical condition medicine.

Brain damage due to stroke triggers a number of pathophysiological reactions, which are based on the accumulation of glutamate with the development of excitotoxicity. The effect of glutamate on NMDA receptors is one of the main factors of neurodegenerative disorders.

Xenon is an anesthetic whose neuroprotective properties have been shown in many experimental studies. However, the clinical part is still presented rather modestly. After it was discovered that xenon is an inhibitor of NMDA receptors, it was shown that xenon can protect neuronal cell cultures from damage caused by NMDA, glutamate, or oxygen-glucose deprivation. It has been experimentally established that xenon is an inhibitor of tissue plasminogen activator (tPA) and dose-dependent inhibits tPA-induced thrombolysis; xenon inhalation after ischemia and reperfusion suppresses ischemic brain damage and tPA-induced cerebral hemorrhages, and damage to the blood-brain barrier.

Exposure to xenon after transient ischemia in rats leads to a decrease in the volume of infarction, depending on the concentration, exposure time and improvement of neurological function 7 days after ischemia. To date, a role has been discovered in the implementation of molecular mechanisms of xenon neuroprotection of double-pore potassium channels (TREK-1), which provide a basic ion current that weakens neuronal excitability, thereby protecting neurons from damage. The role of adenosine triphosphate (ATP)-sensitive potassium channels of the plasmalemma in the realization of the protective properties of xenon is also discussed in the scientific literature. It was shown that under in vitro conditions in the culture of neurons, xenon protected them from damage caused by glucose and oxygen deprivation by activating ATP-sensitive potassium channels in the plasmalemma. There is evidence of the effect of xenon inhalation on the phosphorylation of glycogen synthase-3ß, a key enzyme of the anti-apoptotic neuronal cascade, and an increase in the pool of enzymes involved in the antioxidant protection of the brain. An experimental study showed a distinct anti-inflammatory effect of this anesthetic, which consisted in an increase in the ability of neutrophils to spontaneous apoptosis and a decrease in the expression of adhesion molecules CD11b and CD66b on their surface after modeling an inflammatory reaction. Also, the anti-inflammatory properties of xenon were shown when modeling traumatic brain injury in vivo, when its exposure for 60 minutes caused a significant decrease in the expression of pro-inflammatory genes NF-kB1 and NF-kB2, responsible for the synthesis of cytokines and other molecules involved in inflammation. Considering that the inflammatory reaction that forms in the first hours of ischemic brain damage largely determines the severity of its further course, such an effect on neutrophils can reduce the severity of damage to nervous tissue.

The most interesting is a randomized controlled trial performed by R. Laitio et al. (2016), in which the use of xenon in combination with hypothermia in clinical practice was studied for the first time. In patients who have undergone community-acquired cardiac arrest, xenon inhalation at a concentration of 40 vol.% within 24 hours in combination with hypothermia, led to less damage to the white matter of the brain than with patients using hypothermia alone. The 6-month mortality rate was 27% in the xenon and hypothermia group and 35% in the hypothermia group. However, the study was not powerful enough.

It is important to note that today, despite a large pool of convincing preclinical studies proving the neuroprotective properties of xenon, there is not a single clinical study of its use in ischemic stroke.

Therefore, the research objectives is to determine whether the strategy of using xenon-oxygen mixture inhalation is better than oxygen-air mixture inhalation with respect to the change in scores on the NIHSS, Rankin and Glasgow coma scales on day 7, the duration of stay in the ICU and the frequency of nosocomial pneumonia.

ELIGIBILITY:
Inclusion Criteria:

* Age > 18;
* Ischemic stroke with a NIHSS score at the time of hospitalization from 5 to 15 points
* Score on the Glasgow coma scale ≥ 13 points
* Assessment of the patient no later than 8 hours after the appearance of the first signs of ONMC
* Signed voluntary informed consent to participate in the study.

Exclusion Criteria:

* Myocardial infarction in the previous 6 months
* Body mass index > 35 kg/m2
* Class of chronic kidney disease ≥ 3b
* NYHA class ≥ 3
* Decompensated insulin-dependent diabetes mellitus
* The need for inotropic and/or vasopressor support
* The presence of thrombolysis associated with an actual ischemic stroke
* Documented pneumonia within 3 months before randomization

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 40 (Actual)
Dates: Start 2022-01-01 (Actual); Primary Completion 2024-01-15 (Actual); Study Completion 2024-01-15 (Actual)

PRIMARY OUTCOMES:
National Institutes of Health Stroke Scale | 7 day
  Change of scores on the National Institutes of Health Stroke Scale. Minimal score equal 0. Maximal score equal 42. Less score means better outcome.

SECONDARY OUTCOMES:
Rankin scale | day 7
  Change in Rankin scale scores Minimal score equal 0. Maximal score equal 5. Less score means better outcome.
Glasgow coma scale | day 7
  Change of points on the Glasgow coma scale Minimal score equal 0. Maximal score equal 15. Less score means worse outcome.
Duration of stay in the intensive care unit | 28 days
  day of the intensive care unit discharge - day of the randomization
Nosocomial pneumonia | 28 days
  The incidence of nosocomial pneumonia
Mortality | 28 days
  All cause mortality

CONTACTS AND LOCATIONS:
Overall Officials: Oleg Grebenchikov, MD, Principal Investigator — Negovsky Research Reanimatology Institute
Locations (1):
- V.A. Negovsky Research Institute of General Reanimatology, Federal Research and Clinical Center of Intensive Care Medicine and Rehabilitology, Moscow, Russia

IPD SHARING:
Plan to Share IPD: No